CLINICAL TRIAL: NCT02994446
Title: Saline-Enhanced Radiofrequency (SERF) Catheter Ablation for the Treatment of Ventricular Tachycardia
Acronym: SERF-VT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thermedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD-14-001P
Record Dates: First submitted 2016-12-11; First posted 2016-12-15 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Tachycardia, Ventricular
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SERF Catheter Ablation (Experimental): Ablation of ventricular tachycardia with a saline-enhanced radiofrequency ablation catheter
  Interventions: Device: Saline-Enhanced Radiofrequency Catheter and Ablation System

INTERVENTIONS:
Device: Saline-Enhanced Radiofrequency Catheter and Ablation System — Ablation of ventricular tachycardia with a saline-enhanced radiofrequency ablation catheter
  Other Names: SERF Ablation System and Durablate™ Ablation Catheter

SUMMARY:
The purpose of this study is to demonstrate the technical feasibility of the SERF Catheter and SERF Cardiac Ablation System to eliminate or control ventricular tachycardia (VT)

ELIGIBILITY:
Inclusion Criteria

1. Patient has recurrent, symptomatic, monomorphic VT
2. Patient has drug refractory or drug intolerant VT following use of at least one Class III antiarrhythmic as demonstrated by a recurrent arrhythmia and is not a suitable candidate per the investigator's expert opinion for ongoing or alternative drug therapy
3. A prior failed ablation as evidenced by ICD device therapy within the prior 6 months.
4. Patient has minimum 3 month ICD interrogation history available for evaluation
5. Patient has LVEF > 20%, confirmed by echo or comparable technique during baseline evaluation
6. Patient is at least 18 years old
7. Patient has signed the informed consent, and is willing and able to participate in all study procedures and follow up requirements

Exclusion Criteria

1. Patients with idiopathic VT
2. Patients with VT with ECG or MRI/CT findings suggestive of right ventricular free wall origin findings.
3. Patients with VTs of septal origin may be excluded as such ablations require special care to minimize the risk of heart block, particularly within 2 cm of the AV node/proximal conduction system. Patients requiring ablation at such locations should only be included when the arrhythmia itself is life-threatening or otherwise sufficiently severe to justify the risk.
4. Patient with myocardial infarction (MI) or unstable angina within previous 60 days
5. Patient with cardiac surgery or percutaneous coronary intervention (PCI) within previous 60 days
6. Patient with class IV (NYHA) heart failure
7. Patient with mechanical mitral valve, severe aortic stenosis or flail mitral leaflet
8. Patient with left ventricular assist device planned or required for the procedure
9. Patients with co-morbidities such that they have less than 1 year life expectancy
10. Patient with significant intracardiac and/or laminated thrombus evident by transesophogeal echo (TEE) or transthoracic echo (TTE) (with contrast) within 2 days of the ablation procedure
11. Patient with thrombocytopenia or other coagulopathy
12. Women who are or may potentially be pregnant. (must be post-menopausal or have a negative pregnancy test)
13. Patient with other acute illness or active systemic infection (unrelated to VT or its origin)
14. Significant congenital anomaly heart disease or anomaly
15. Allergy or contraindications to the medications/agents used during a standard ablation/EP intervention.
16. Patient concurrently enrolled in any other investigational drug or device study that the investigator deems would interfere with study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Events that are potentially device-related | Within 30 days of ablation
Major Adverse Cardiac Events | Within 2 days after ablation procedure
  MACE will be accessed from time of ablation to time of discharge from hospital following the ablation (generally within 2 days of ablation procedure).
Non-inducibility of clinical ventricular tachycardia (VT) and/or elimination of clinically relevant scar or channels | At completion of ablation procedure

SECONDARY OUTCOMES:
Intraprocedural non-inducibility and/or scar homogenization of target VT | At completion of ablation procedure
Elimination of the target VT and/or reduction in number of VT episodes | Within first 6 months of ablation procedure

CONTACTS AND LOCATIONS:
Overall Officials: Douglas L. Packer, MD, Study Director — Mayo Clinic; Atul Verma, MD, Principal Investigator — Southlake Regional Health Centre
Locations (3):
- Canada (3):
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Montreal Heart Institute - Institut de Cardiologie de Montréal, Montreal, Quebec
  - Quebec Heart and Lung Institute - Institut universitaire de cardiologie et de pneumologie de Québec, Québec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Packer DL, Wilber DJ, Kapa S, Dyrda K, Nault I, Killu AM, Kanagasundram A, Richardson T, Stevenson W, Verma A, Curley M; SERF Investigators. Ablation of Refractory Ventricular Tachycardia Using Intramyocardial Needle Delivered Heated Saline-Enhanced Radiofrequency Energy: A First-in-Man Feasibility Trial. Circ Arrhythm Electrophysiol. 2022 Aug;15(8):e010347. doi: 10.1161/CIRCEP.121.010347. Epub 2022 Jul 1. PMID 35776711